CLINICAL TRIAL: NCT06058143
Title: Efficacy of Crenel Lateral Interbody Fusion Combined With Lateral Plate Fixation Versus Transforaminal Lumber Interbody Fusion for Lumbar Spinal Stenosis Combined With Lumbar Instability
Brief Title: Crenel Lateral Interbody Fusion Combined With Lateral Plate Fixation for LSS Combined With Lumbar Instability
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mars515
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Lumbar Spinal Stenosis; Lumbar Instability
Keywords: lumbar spinal stenosis;lumbar instability
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Patients who received CLIF-LP treatment
  Interventions: Procedure: CLIF-LP
- Group 2 (Active Comparator): Patients who received TLIF treatment
  Interventions: Procedure: TLIF

INTERVENTIONS:
Procedure: CLIF-LP — CLIF-LP surgery method was applied
  Arms: Group 1
Procedure: TLIF — TLIF surgery method was applied
  Arms: Group 2

SUMMARY:
At present, interbody fusion is the mainstream treatment for patients with lumbar spinal stenosis (LSS) and lumbar instability. However, the choice of interbody fusion for LSS patients with lumbar instability remains controversial. Recently, we developed crenel lateral interbody fusion combined with lateral plate fixation(CLIF - LP) for patients with LSS and lumbar instability. This surgical method has many advantages and showed good results for patients with LSS and lumbar instability. Therefore, we propose the following hypothesis: The clinical and imaging efficacy of CLIF-LP in the treatment of LSS patients with lumbar instability is not inferior to that of traditional transforaminal lumber interbody fusion (TLIF).

DETAILED DESCRIPTION:
At present, interbody fusion is the mainstream treatment for patients with lumbar spinal stenosis (LSS) and lumbar instability. However, the choice of interbody fusion for LSS patients with lumbar instability remains controversial. Recently, we developed crenel lateral interbody fusion combined with lateral plate fixation(CLIF - LP) for patients with LSS and lumbar instability. This surgical method has the advantages of direct view operation, "safe" psoas major approach, application of modified retractor, and lateral plate reinforcement, which not only significantly improves the postoperative lumbar function and nerve function of patients with LSS and lumbar instability, but also significantly reduces related complications, accelerates rehabilitation, and reduces the medical cost of patients.

Therefore, we propose the following hypothesis: The clinical and imaging efficacy of CLIF-LP in the treatment of LSS patients with lumbar instability is not inferior to that of traditional transforaminal lumber interbody fusion (TLIF).

ELIGIBILITY:
Inclusion Criteria:

1. Age 50-80 years old
2. Patients diagnosed with clinical symptoms of lumbar spinal stenosis, neurogenic intermittent claudication, the patient's walking ability is highly limited, and the quality of life is severely reduced
3. Imaging diagnosis of 1-2 LSS patients, consistent with clinical symptoms
4. Lumbar spine instability can be considered if one of the following three criteria is met: ① mechanical back pain with severe (VAS > 7) (pain aggravates with weight bearing). Radiographs of lumbar hyperextension and flexion show a slip of at least 3mm between the two vertebrae, or a rotation Angle of 11°. ③ Degenerative slip
5. Formal conservative treatment is ineffective for more than 3 months
6. No history of lumbar surgery
7. American College of Physicians ASA Grade I or II
8. Subjects voluntarily sign informed consent as subjects

Exclusion Criteria:

1. In patients with significant symptoms of lumbar radiculopathy, the pain from postural changes cannot be relieved
2. Bone stenosis, including developmental lumbar spinal stenosis
3. Free nucleus pulposus tissue into the spinal canal or cause spinal canal compression of the small joint cyst
4. Patients with hypertrophy of the yellow ligament or small joint cyst as the main pressure
5. Intervertebral space or posterior facet joints have fused
6. Infectious, traumatic and neoplastic diseases of the lumbar spine
7. Patients who are unable to undergo MRI
8. Some medical conditions, such as metabolic bone disease, autoimmune disease, poliomyelitis sequelae, osteoporosis, history of poor bone healing, and long-term oral steroids, were determined by the investigators to be unsuitable for inclusion in the study
9. Patients with evidence of neurological disorders (such as peripheral neuropathy), neuromuscular disorders (such as multiple sclerosis, Parkinson's disease, etc.), or systemic diseases (such as inflammatory arthritis) that affect bodily function
10. The patient has participated in other clinical trials in the past 3 months
11. Patients with poor adherence, judged by the researchers to be unable to complete the trial according to the study plan, such as schizophrenia and dementia, did not provide consent to volunteer to participate in the clinical study

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability index (ODI) | 24 months after surgery
  Lumbar function was assessed by the Oswestry Disability index (ODI) at 24 months after surgery. ODI includes 10 items, including waist and leg pain, personal life care, lifting heavy objects, walking, sitting, standing, sleeping, sexual life, social life, and whether you can travel freely. The total score is 50 points, and the lower the score, the better the function of the lumbar spine.

SECONDARY OUTCOMES:
Visual analogue scale（VAS） | 1 month, 3 months, 6 months, 12 months and 24 months after surgery
  Visual analogue scale (VAS) was used for pain scores, and mild pain was 0-3 points, which was tolerable; Moderate pain is 4 ~ 6 points, strong pain affects rest, but can be tolerated; Severe pain is a score of 7 to 10, and the patient's pain is intensified and unbearable.
Japanese Orthopaedic Association (JOA) | 1 month, 3 months, 6 months, 12 months and 24 months after surgery
  The JOA lumbar spine score included four aspects: subjective symptoms, clinical signs, daily activities and bladder function. The highest JOA score was 29 and the lowest was 0. The lower the score was, the more severe the symptoms and the more obvious the dysfunction.
EuroQoL-5D-5L | 1 month, 3 months, 6 months, 12 months and 24 months after surgery
  This scale is a multidimensional measure of health-related quality of life, and it is also the most widely used universal utility scale. EQ-5D-5L consists of five dimensions, namely mobility, self-care, daily activities, pain or discomfort, anxiety or depression, each area is rated on a five-point scale (i.e., no problem, mild problem, moderate problem, severe problem, extreme problem), with higher scores indicating worse conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Ning Zhang, PhD, Study Director — Second Affiliated Hospital, School of Medicine, Zhejiang University

IPD SHARING:
Plan to Share IPD: No